CLINICAL TRIAL: NCT00242853
Title: An Enabling Study to Investigate the Correlation of Biomarkers of the Activity of Inducible Nitric Oxide Synthase (iNOS) With Disease Activity and Treatment Response in Patients With Rheumatoid Arthritis(RA)
Brief Title: A Study To Investigate Markers Of Inflammation In Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: RA4102651
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis
Keywords: iNOS; Rheumatoid arthritis; Exhaled NO
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Power doppler ultrasonography
Procedure: High frequency ultrasonography
  Other Names: Exhaled nitric oxide assessment; Power doppler ultrasonography
Procedure: Exhaled nitric oxide assessment

SUMMARY:
This study is being conducted to validate various biomarkers in patients with RA with varying levels of disease severity. Subjects with a diagnosis of rheumatoid arthritis (RA) will be included as controls. The sudy will measure the baseline levels and the intra- and inter-subject variability of exhaled nitric oxide (NO) in patients with inactive/mild and moderate/severe RA on stable therapy or during a course glucocorticoids. In addition exhaled NO levels will be correlated with intra-articular inflammation (power Doppler ultrasonography) as well as markers of systemic inflammation (CRP, ESR).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of rheumatoid or osteo-arthritis.
* Weight greater than 45kg (females) or 50kg (males) but not overweight.
* Non-smokers.
* Taking stable anti-inflammatory medication for Rheumatoid Arthritis (RA) or Osteoarthritis (OA) for at least 8 weeks.

Exclusion criteria:

* Taking regular doses of glucocorticoid medication (greater than 5mg/day).
* Currently taking biological treatment for RA.
* Recent participation in another clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom